CLINICAL TRIAL: NCT04927286
Title: Implementing Learning 2 BREATHE in Campus Connections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008
Record Dates: First submitted 2021-06-03; First posted 2021-06-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Mindfulness
Keywords: adolescents; mindfulness; ecological momentary assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentoring+Mindfulness (Experimental)
  Interventions: Behavioral: Learning to Breathe
- Mentoring as usual (Active Comparator)
  Interventions: Behavioral: Campus Connections

INTERVENTIONS:
Behavioral: Learning to Breathe — Learning to Breathe is an evidence-based mindfulness curriculum for adolescents
  Arms: Mentoring+Mindfulness
Behavioral: Campus Connections — Campus Connections is a mentoring program for at-risk adolescents
  Arms: Mentoring as usual

SUMMARY:
The overall objective of this study is to investigate a mindfulness-based intervention's feasibility/acceptability and effectiveness for improving eating behaviors and depression symptoms among adolescents (9-18y; 63% living on low-income), referred to a community-based mentoring program for being "at-risk for not reaching their full potential" (e.g., Department of Human Services involvement, behavioral/emotion problems). As a part of this study, we will also characterize the real-time relationships among life stressors, untrained state mindfulness, and emotion regulation difficulties in adolescents' daily lives and determine to what extent an MBI helps adolescents to maintain mindfulness and emotion regulation in moments when they experience a stressor.

ELIGIBILITY:
Inclusion Criteria:

* Mentees (adolescents) participating in campus connections who are 9-18y and English speaking

Exclusion Criteria:

* Mentees (adolescents) that are not participating in campus connections

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Reward-based Eating Behaviors | Through study completion, an average of 6 months
  Changes in Reward-based eating behaviors for all participants will be assessed with the Reward-based eating behaviors scale (Mason et al., 2017)
Internalizing and Externalizing Symptoms | Through study completion, an average of 6 months
  The Brief problem monitor (Achenbach et al., 2011) will be used to assess for changes in internalizing (e.g., depression symptoms) and externalizing symptoms for all participants.
Mindfulness | Through study completion, an average of 6 months
  The mindfulness attention and awareness scale (Brown & Ryan, 2003) will be used to assess for changes in mindfulness for all participants
Emotion Regulation | Through study completion, an average of 6 months
  The Difficulties in Emotion Regulation Scale-Short Form (Kaufman et al., 2016) will be used to assess for changes in difficulties with emotion regulation for all participants

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State Univeristy, Fort Collins, Colorado, United States

REFERENCES:
- [Derived] Miller-Chagnon RL, Shomaker LB, Prince MA, Krause JT, Rzonca A, Haddock SA, Zimmerman TS, Lavender JM, Sibinga E, Lucas-Thompson RG. The benefits of mindfulness training for momentary mindfulness and emotion regulation: A randomized controlled trial for adolescents exposed to chronic stressors. J Consult Clin Psychol. 2024 Dec;92(12):800-813. doi: 10.1037/ccp0000910. PMID 39715423
- [Derived] Miller RL, Shomaker LB, Prince MA, Haddock S, Rzonca A, Krause JT, Zimmerman T, Lavender JM, Sibinga E, Lucas-Thompson RG. Momentary effects of life stressors on mindfulness and emotion regulation difficulties among adolescents exposed to chronic stressors. Stress Health. 2024 Oct;40(5):e3414. doi: 10.1002/smi.3414. Epub 2024 Apr 29. PMID 38685855